CLINICAL TRIAL: NCT05988229
Title: Tools to Improve Discharge Equity (TIDE) at Hospital Discharge for Patients With Limited English Proficiency: A Randomized Controlled Trial
Brief Title: Tools to Improve Discharge Equity (TIDE) Pilot RCT
Acronym: TIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-43873
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hospital Discharge
Keywords: Limited English proficiency; Hospital Discharge Teaching; Spanish speaking; Haitian Creole speaking; Cape Verdean Creole speaking; Vietnamese speaking

STUDY DESIGN:
Intervention Model Description: Block randomization stratified by language and level of care (observation unit versus inpatient floor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discharge equity tools (Experimental): Participants randomized into this arn will receive the toolkit of linguistically appropriate discharge teaching aids at hospital discharge.
  Interventions: Other: Toolkit to improve discharge equity
- Standard of hospital discharge care (No Intervention): Participants randomized into this arm will receive the standard of care at hospital discharge.

INTERVENTIONS:
Other: Toolkit to improve discharge equity — Linguistically appropriate discharge teaching aids: a medication calendar, pictographics added to the after visit summary (AVS), and an audio recording of the discharge teaching.
  Arms: Discharge equity tools

SUMMARY:
The investigators will test the impact of a package of linguistically appropriate discharge teaching tools against current standard of care for patients with Limited English proficiency (LEP) in an unblinded randomized controlled trial. The tools include an expanded medication calendar in English and the patients' preferred language, pictographics to illustrate return precautions (what signs/symptoms require further evaluation), an audio recording of the nurse reviewing the After Visit Summary (composed by providers) to allow for review by patients and caretakers after discharge.

The investigators will evaluate the effectiveness of the package of discharge teaching tools on patients' understanding/recall, key implementation outcomes, and secondary clinical outcomes via a structured interview 1-2 weeks after discharge and chart review 30 days after discharge.

The objectives of this research study are:

1. test the effectiveness of a linguistically appropriate toolkit for improving patient understanding of discharge instruction content
2. Assess the feasibility and fidelity of the intervention in anticipation of a multi-site implementation trial
3. assess the feasibility and appropriateness of the linguistically appropriate toolkit to nurses and in-person interpreters
4. to assess the acceptability of the intervention to patients and their satisfaction with it
5. to collect data on implementation context in anticipation for a multi-site trial
6. to collect preliminary data on the toolkit's impact on clinical outcomes including medication adherence and hospital re-utilization.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Labeled in medical record as preferring one of the following four languages: Spanish, Haitian Creole, Cape Verdean Creole, or Vietnamese
* Admitted to medicine team at BMC
* Age 18 years or older
* Being discharged home (to the community)
* Admitted to Boston Medical Center (BMC) hospital units (Menino 7 East, 7 West, and Menino Observation)

Nurses and Interpreters

* Caring for patient enrolled in trial

Family/Visitors

* Present at time of discharge for patient enrolled in trial

Exclusion Criteria:

Patients

* On airborne infections precautions
* On clostridium difficile (C diff) precautions
* On suicide precautions
* Nurse report of participant displaying cognitive impairment, delirium, or aggression
* Enrolled in trial during a prior admission

Nurses and Interpreters

* None

Family/Visitors

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Patient understanding of discharge instructions | 1-2 weeks post discharge
  Assessed by a composite score of six key domains of discharge instructions (primary diagnosis, self-care instructions, return precautions, medication changes, medication indications, follow-up) as determined by two physician adjudicators (1=poor, 4 = near perfect). Higher scores demonstrate better understanding.
Patient understanding of primary diagnosis of hospitalization | 1-2 weeks post discharge
  Determined by two physician adjudicators (1=poor, 4 = near perfect). Higher scores demonstrate better understanding.

SECONDARY OUTCOMES:
Implementation effectiveness | 18 months
  Effectiveness will be assessed by observations of and comments from patients, nurses and visitors from qualitative interviews related to the adoption, acceptability, appropriateness, and feasibility of the discharge process
Hospital re-utilization | 30 days
  Assessed by a combined outcome of admission or emergency department (ED) visit within 30 days of index discharge
Number of participants with completion of primary care follow-up | 30 days
  Assessed from participants' medical records
Participant participation in discharge teaching | 1-2 weeks
  Participants are observed by a research team member during discharge teaching and will document the number of questions asked.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Austad, MD MPH, Principal Investigator — Boston Medical Center, Family Medicine
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Austad K, Thai C, Zavatti A, Nguyen N, Bautista-Hurtado D, Kenney P, Lugo N, Lee JH, Lanney H, Xuan Z, Cordova-Ramos EG, Drainoni ML, Jack B. Tools to improve discharge equity: Protocol for the pilot TIDE trial. Contemp Clin Trials Commun. 2024 Dec 21;43:101419. doi: 10.1016/j.conctc.2024.101419. eCollection 2025 Feb. PMID 39810841